CLINICAL TRIAL: NCT06543849
Title: The Impact of Targeted Temperature Management Duration on Thrombin Function in Cardiac Arrest Patients (ITTC Trial): A Single-Center, Prospective, Randomized Controlled Trial
Brief Title: The Impact of Targeted Temperature Management Duration on Thrombin Function in Cardiac Arrest Patients
Acronym: ITTC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-1-26-5
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Targeted Temperature Management; Cardiac Arrest; Thrombin Function; Treatment Duration
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-hour treatment (Sham Comparator)
  Interventions: Procedure: Target Temperature Management Treatment
- 72-hour treatment (Active Comparator)
  Interventions: Procedure: Target Temperature Management Treatment

INTERVENTIONS:
Procedure: Target Temperature Management Treatment — Target Temperature Management Treatment

SUMMARY:
This study will be a single-center, prospective, randomized controlled trial with an estimated sample size of 64 patients. Eligible patients will be randomly assigned in a 1:1 ratio to receive TTM for either 24 hours or 72 hours. The primary outcome measure will be the changes in thrombin function indices at various time points during TTM treatment in both groups. The secondary endpoints of the study include additional coagulation function indicators, the incidence of bleeding-related events between the two groups, the amount of blood products used, the incidence of thrombotic events, and the CPC scores at 28 days and 6 months for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years;
2. Glasgow Coma Scale score of less than 8 upon admission;
3. patients resuscitated after out-of-hospital cardiac arrest; and (4) patient or their legal representative has signed the informed consent form.

Exclusion Criteria:

1. cardiac arrest caused by irreversible factors such as trauma or poisoning;
2. cardiac arrest due to terminal conditions like advanced cancer;
3. uncorrected persistent cardiogenic shock, defined as a systolic blood pressure below 90 mmHg despite treatment with fluid resuscitation, vasopressors, and inotropic agents;
4. pre-existing cerebrovascular disease or CT-confirmed intracerebral hemorrhage upon admission;
5. pre-arrest Cerebral Performance Category (CPC) score between 3 and 5;
6. bradycardia or sick sinus syndrome following the return of spontaneous circulation;
7. pre-existing coagulation disorders or severe bleeding tendencies;
8. pregnant or breastfeeding women, or women of childbearing age with elevated serum hCG levels;
9. presence of treatment limitations (such as refusal by the patient or legal representative to undergo advanced life support, including mechanical ventilation, chest compressions, or targeted temperature management);
10. determination by the principal investigator that the patient is unsuitable for the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prothrombin Time (PT) | 4 days
  The primary outcome measure is the statistical differences in prothrombin time (PT) between the two groups of patients at various time points.
Prothrombin Activity (PA) | 4 days
  The primary outcome measure is the statistical differences in prothrombin activity (PA) between the two groups of patients at various time points.
Activated Partial Thromboplastin Time (APTT) | 4 days
  The primary outcome measure is the statistical differences in activated partial thromboplastin time (APTT) between the two groups of patients at various time points.
Thrombin Time (TT) | 4 days
  The primary outcome measure is the statistical differences in thrombin time (TT) between the two groups of patients at various time points.

SECONDARY OUTCOMES:
The concentration of D-dimer (D-D) | 4 days
  The primary outcome measure is the statistical differences in D-dimer (D-D) between the two groups of patients at various time points.
International Normalized Ratio (INR) | 4 days
  The primary outcome measure is the statistical differences in international normalized ratio (INR) between the two groups of patients at various time points.
The concentration of plasmin-α2-plasmin inhibitor complex (PIC) | 4 days
  The primary outcome measure is the statistical differences in plasmin-α2-plasmin inhibitor complex (PIC) between the two groups of patients at various time points.
The concentration of fibrinogen (FBG) | 4 days
  The primary outcome measure is the statistical differences in fibrinogen (FBG) between the two groups of patients at various time points.
The concentration of thrombin-antithrombin complex (TAT) | 4 days
  The primary outcome measure is the statistical differences in thrombin-antithrombin complex (TAT) between the two groups of patients at various time points.
The concentration of thrombomodulin (TM) | 4 days
  The primary outcome measure is the statistical differences in thrombomodulin (TM) between the two groups of patients at various time points.
The concentration of tissue-type plasminogen activator inhibitor complex (T-PAIC) | 4 days
  The primary outcome measure is the statistical differences in tissue-type plasminogen activator inhibitor complex (T-PAIC) between the two groups of patients at various time points.
thrombelastogram (TEG) | 4 days
  The primary outcome measure is the statistical differences in thrombelastogram (TEG) between the two groups of patients at various time points.
Platelet Count (PLT) | 4 days
  The primary outcome measure is the statistical differences in platelet count (PLT) between the two groups of patients at various time points.
The rate of bleeding-related events | 4 days
  The incidence of bleeding-related events in the two groups of patients, including gastric occult blood, fecal occult blood, intracerebral hemorrhage, or bleeding in other organs.
The Milliliters of blood products | 4 days
  The usage of blood products, including red blood cells, platelets, and fresh frozen plasma.
CPC Score | 28 days and 6 months
  CPC = Cerebral Performance Category Score. The Secondary Outcome of the study is analyzed as the proportion of patients with good neurological outcome in the two groups, (CPC 1-2) at 6 months after CA.

OTHER OUTCOMES:
The percentage of serious adverse events during the 4-day treatment period | 4 days
  The primary safety measure is the percentage of serious adverse events during the 4-day treatment period, including any events that cause permanent damage to organs, are life-threatening, or result in death.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors